# Statistical Analysis Plan

## Viromed Co., Ltd

US 06-1-001

# A Phase I, Dose-Escalation, Single Center Study to Assess the Safety and Tolerability of VM202 in Subjects with Critical Limb Ischemia

# Protocol Version 5.0- November 29, 2007

Sponsor:

Prepared by:

Version: 2

Date of Creation: September 14, 2007

Last Updated: January 10, 2008

# TABLE OF CONTENTS

| LIS | T OF | ABBREVIATIONS | 4 |
|-----|-------|-------------------------------------------|------|
| DE | FINIT | IONS | 6 |
| 1. | INTE | RODUCTION | 7 |
| 2. | OBJ | ECTIVES | 7 |
| | 2.1 | PRIMARY OBJECTIVE | |
| | 2.2 | SECONDARY OBJECTIVES | |
| 3. | STU | DY OVERVIEW | 7 |
| 4. | | ERAL ANALYSIS CONSIDERATIONS | |
| 5. | ANA | LYSIS POPULATIONS | 9 |
| 6. | SUB. | JECT DISPOSITION | 9 |
| 7. | DEM | OGRAPHIC AND BASELINE CHARACTERISTICS | 9 |
| 8. | EFFI | CACY ANALYSES | 9 |
| | 8.1 | EFFICACY VARIABLES | 9 |
| | 8.2 | BASELINE VALUES | 10 |
| | 8.3 | HANDLING MISSING DATA | 10 |
| | 8.4 | INTERIM ANALYSES | 10 |
| | 8.5 | MULTIPLICITY ADJUSTMENTS | |
| | 8.6 | By Center Analyses | 10 |
| 9. | MET | THODS OF EFFICACY ANALYSIS | 10 |
| | 9.1 | AREA OF ISCHEMIC ULCER | 10 |
| | 9.2 | HEMODYNAMIC ASSESSMENTS | 11 |
| | 9.3 | VISUAL ANALOGUE SCALE FOR PAIN | 11 |
| | 9.4 | TRANSCUTANEOUS OXYGEN PRESSURE ASSESSMENT | 11 |
| | 9.5 | SUBJECT ANALGESIC USE | 11 |
| | 9.6 | HIGH RESOLUTION MRA | 12 |
| 10. | SAFI | ETY ANALYSES | 12 |
| | 10.1 | STUDY DRUG EXPOSURE | 12 |
| | 10.2 | ADVERSE EVENTS | 12 |
| | 10.3 | CLINICAL LABORATORY EVALUATION | 13 |
| | 10.4 | PHYSICAL EXAMINATIONS | 13 |
| | | VITAL SIGNS | |
| | 10.6 | RETINAL FUNDOSCOPY | 14 |
| | 10.7 | INFECTION TESTS | 14 |
| | 10.8 | Tumor Marker | 14 |
| | 10.9 | INJECTION SITE REACTION | 14 |
| | 10.10 | PRIOR AND CONCOMITANT MEDICATIONS | . 14 |

| 11. PHARMACOKINETICS | 15 |
|-----------------------------------------|----|
| 12. PHARMACODYNAMICS | 15 |
| APPENDIX A: LIST OF TABLES AND LISTINGS | 16 |
| APPENDIX B: TABLE LAYOUTS | 20 |

#### LIST OF ABBREVIATIONS

ABI ankle-brachial index

AE adverse event

ALT alanine transaminase (SGPT)
AST aspartate transaminase (SGOT)

AUC area under the plasma concentration time curve

BUN blood urea nitrogen
°C degrees Celsius
CBC complete blood count

cDNA complementary deoxyribonucleic acid

CHF congestive heart failure
CFR Code of Federal Regulation
CLI critical limb ischemia

Cm centimeter(s)

C<sub>max</sub> maximum concentration of drug

CRF case report form

CRO clinical research organization

CVD cardiovascular disease

D day(s) dL deciliter(s)

DSMC Data Safety Monitoring Committee

ECG electrocardiogram

ET endothelin

°F degrees Fahrenheit

FDA Food and Drug Administration

G gram(s)

GCP Good Clinical Practices HGF hepatocyte growth factor

IBC Institutional Biosafety Committee

ICH International Conference on Harmonisation IDUR investigational drug utilization record

IND Investigational New Drug
INR international normalized ratio
IRB Institutional Review Board

IV intravenous

IVRS Interactive Voice Response System

Kg kilogram(s)

LOCF last observation carried forward

## LIST OF ABBREVIATIONS (CONTINUED)

LV left ventricular Mg milligram(s) Min minute(s)

mmHg millimeters mercury

MRA magnetic resonance angiography

MTD maximum tolerated dose

N number Ng nanogram(s)

NIH National Institutes of Health NYHA New York Heart Association

 $O_2$  oxygen

OBA Office of Biotechnology Activities

PAD peripheral artery disease
pH hydrogen ion concentration
PHI protected health information

PPG photoplethysmograph

PTA percutaneous transluminal angioplasty

QD once daily
RBC red blood count
SAE serious adverse event
SAP Statistical Analysis Plan

sDBP sitting diastolic blood pressure

SE standard error

SGPT serum glutamic pyruvic transaminase (same as ALT)

SOC System Organ Class

SVR systemic vascular resistance

t<sub>1/2</sub> elimination half-life

time of occurrence for maximum (peak) drug concentration

TBI toe-brachial index

TcPO<sub>2</sub> Transcutaneous Oxygen Pressure Assessment

VAS visual analog scale

VEGF vascular endothelial growth factor

vs. versus

WBC white blood count

WHO World Health Organization

## **DEFINITIONS**

Adverse Event An adverse event (AE) is the development of an undesirable

medical condition following or during exposure to a

pharmaceutical product, whether or not considered causally

related to the product.

Baseline The last non-missing value prior to first dose of study drug. Serious AE An AE occurring at any dose that: results in death; is a

life-threatening experience; requires hospitalization or prolongation of an existing hospitalization; results in a persistent or significant disability/incapacity; or is a

congenital anomaly/birth defect in the offspring of a subject

who received study drug.

Treatment-emergent AE AEs with an onset time after the initial dose of study drug.

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of ViroMed Co., Ltd. Protocol US 06-1-001 [A Phase I, Dose-Escalation, Single Center Study to Assess the Safety and Tolerability of VM202 in Subjects with Critical Limb Ischemia]. The purpose of this plan is to provide specific guidelines from which the analysis will proceed. Any deviations from these guidelines will be documented in the clinical study report (CSR).

## 2. OBJECTIVES

## 2.1 Primary Objective

The primary objective of this study is to evaluate the safety and tolerability of intramuscular VM202 as a vehicle for therapeutic angiogenesis in subjects with critical limb ischemia.

## 2.2 Secondary Objectives

The secondary objectives of the study will include the following exploratory evaluations:

- To investigate the effects of the intramuscular VM202 to improve pain at rest and/or to heal ischemic ulcers of the affected limb. The VAS assessment tool will be used for this evaluation:
- To evaluate the anatomic and physiological extent of collateral vessel development in subjects with critical limb ischemia as measured by MRA;
- To evaluate the change in serum HGF levels from Day 1 to Day 59;
- To evaluate the change in VM202 DNA levels from Day 1 to Day 59;
- To evaluate the immune response to HGF in subjects with CLI as measured by the change in anti-HGF antibodies from Day 1;
- To evaluate the ability of VM202 to stimulate endothelial progenitor cells as measured by the change in endothelial cell progenitor assay levels from screening to Day 59.

## 3. STUDY OVERVIEW

This is a prospective, dose-escalation single center study to evaluate the safety and tolerability of intramuscular VM202 in subjects with critical limb ischemia.

Subjects selected for this study will have critical limb ischemia that has not responded to standard therapy with symptoms including pain at rest or ischemic ulcers.

The study will consist of four (4) cohorts with a total of 3 subjects enrolled in each cohort to VM202. The cohorts will be based on the planned different amounts of VM202 to be given. Planned levels of VM202 to be administered (defining the 4 cohorts) are the following: 2 mg, 4 mg, 8 mg and 16 mg. For each dose cohort, VM202 will be administered as a local intramuscular injection in 2 divided doses with a 2-week interval between the injections. Preliminary efficacy (hemodynamic assessments), safety and tolerability will be evaluated at Baseline (screening) and at designated time points throughout the study.

After all subjects in the first dose cohort have completed the 30-day ( $\pm 2$  days) follow-up visit following the 1st dose of study drug, an interim safety evaluation will be performed with the submission of safety data to the Data Safety Monitoring Committee (DSMC). If the DSMC recommends continuing the study, the second dose cohort will be treated. This process will be repeated between the second and third dose cohort and between the third and fourth dose cohort. All 4 dose cohorts will be followed for up to five years from the time of the first dose of study drug administration. If a dose limiting toxicity (DLT) is observed in one subject in any dose group, three additional subjects will be added to the dose cohort in which the toxicity was observed. If no additional DLTs are observed in the 6 subjects in this dose level, it will be considered the maximum tolerated dose (MTD). If a DLT occurs in 2/6 subjects, then the preceding dose level will be considered the MTD.

## 4. GENERAL ANALYSIS CONSIDERATIONS

The statistical analyses will be reported using summary tables, figures, and data listings. Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums. Categorical variables will be summarized by counts and by percentage of subjects in corresponding categories.

Individual subject data obtained from the case report forms (CRFs), pharmacokinetic/pharmacodynamic data, and any derived data will be presented by subject in data listings.

All analyses and tabulations will be performed using SAS® Version 8.2 or higher on a PC platform. Tables and listings will be presented in RTF format. Upon completion, all SAS® programs will be validated by an independent programmer. In addition, all program output will undergo a senior level statistical review. The validation process will be used to confirm that statistically valid methods have been implemented and that all data manipulations and calculations are accurate. Checks will be made to ensure accuracy, consistency with this plan, consistency within tables, and consistency between tables and

corresponding data listings. Upon completion of validation and quality review procedures, all documentation will be collected and filed by the project statistician or designee.

## 5. ANALYSIS POPULATIONS

The following subject populations will be used for analysis:

The Safety population will include all subjects who received at least one dose of study drug medication. Safety analysis will be performed on the Safety population.

The Intent-to-Treat (ITT) population will include all subjects who received at least one dose of study drug medication and had at least one post dose assessment. Efficacy, pharmacokinetic (PK) and pharmacodynamic (PD) analysis will be performed on the ITT population.

## 6. SUBJECT DISPOSITION

Subject disposition information will be summarized for all subjects by dose cohort. Summaries will include: the number of enrolled subjects, the number of subjects in each analysis population, the number of subjects who received both planned doses of VM202, the last scheduled visit completed, the number of subjects completing the study and the primary reason for discontinuation.

## 7. DEMOGRAPHIC AND BASELINE CHARACTERISTICS

Demographic variables include: age, sex, ethnicity, race. Medical history and peripheral vascular disease intervention history at baseline will also be considered. Demographic and baseline characteristics will be summarized for the Safety and ITT analysis populations.

#### 8. EFFICACY ANALYSES

Efficacy analysis will be based on the ITT analysis population. The efficacy analysis generated for this study is intended to be used for preliminary and exploratory considerations and is not meant to be confirmatory in nature.

## 8.1 Efficacy Variables

The following efficacy endpoints of equal interest will be collected and analyzed:

- Area of Ischemic Ulcer (largest contiguous area of ulceration)
- Hemodynamic Assessments to include:
  - Ankle-Brachial Index (ABI)

- 2. Toe-Brachial Index (TBI)
- 3. Wave Form Analysis (PVR);
- Pain Visual Analogue Scale (VAS) Score;
- Transcutaneous Oxygen Pressure Assessment (TcPO<sub>2</sub>);
- Subject Analgesic Use;
- High resolution MRA.

## 8.2 Baseline Values

The baseline value for each variable is the value recorded at the last visit on or before start of dosing. In most cases, baseline values are expected to be based on the assessment collected at the Day 1 (Pre-Dose) visit.

## 8.3 Handling Missing Data

Only data collected will be used for analysis. Missing values will not be imputed for this study.

## 8.4 Interim Analyses

No interim analysis of efficacy data is planned.

## 8.5 Multiplicity Adjustments

No alpha adjustments for multiple comparisons will be made since this is an open-label study with no formal cohort comparisons.

## 8.6 By Center Analyses

As this is a single center study, no by-center analysis is planned.

## 9. METHODS OF EFFICACY ANALYSIS

## 9.1 Area of Ischemic Ulcer

For each subject, the ulcer with the largest contiguous area will be measured both before and after the first dose of study medication. Planned post dose measurements of the ulcer include measurements at Day 15 (Pre-Dose), Day 28, Day 59, Day 91, Day 180 and Day 365. Ulcer measurements will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized.

## 9.2 Hemodynamic Assessments

Hemodynamic assessments will be taken before the first dose of medication and at Day 15 (Pre-Dose), Day 28, Day 59, Day 91, Day 180 and Day 365. Hemodynamic assessments will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized. Hemodynamic assessments, all in units of mmHg, include the following:

- Ankle Brachial-Index measurements taken on both legs. Counts and percentages
  of the index limb (right/left) will be also be presented;
- Toe Brachial-Index measurements taken on toe of right and left foot.

Confirmation that wave form analysis (PVR) was collected will be presented in listings.

## 9.3 Visual Analogue Scale for Pain

Throughout the study, subjects will be asked to assess the level of pain they feel by placing a perpendicular line on a scale of 0 (No Pain) to 100 (Pain as bad as it can be). The subject's Visual Analogue Scale (VAS) score will be determined by where the subject places the perpendicular line. Measurements of VAS will be collected prior to first study drug administration and at Day 15 (Pre-Dose), Day 28, Day 59, Day 91, Day 180 and Day 365 of the study. VAS measurements will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized.

## 9.4 Transcutaneous Oxygen Pressure Assessment

Before the first dose of medication and at Day 15 (Pre-Dose), Day 28, Day 59, Day 91, Day 180 and Day 365 of the study, assessments of the transcutaneous oxygen pressure (TcPO<sub>2</sub>) in various regions of the body will be taken. Those regions include assessments of the anterior calf, posterior calf, dorsum foot and chest. TcPO<sub>2</sub> measurements for each body region will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized.

## 9.5 Subject Analgesic Use

Concomitant medication use will be collected throughout the study on an ongoing basis. A review of concomitant medications used by subjects will be carried out to determine which concomitant medications were administered for analgesic use. Based on the review of concomitant medications, subjects will be classified as either having used an analgesic or not. Counts and percentages showing the number of subjects having used or not having used analgesics will be presented.

## 9.6 High Resolution MRA

Occluded arteries will be identified as one of the following categories on CRFs: Super femoral artery (SFA), popliteal, peroneal, anterior tibeal, post tibial, infrapopliteal. Information regarding occluded arteries will be presented in listings. The quantitative blood flow of the target occluded artery and the volumetric analysis of newly developed artery will be not be recorded on the CRF. That information will be in a separate report compiled by the site and another vendor.

## 10. SAFETY ANALYSES

All subjects who received study drug will be included in the safety analyses, analyzed according to the study treatment actually received.

## 10.1 Study Drug Exposure

Study drug exposure will be summarized by dose cohort for Day 1 (planned first dose of VM202) and Day 15 (planned second dose of VM202). Categorical variables to be summarized using counts and percentages include "Was dose administered?" (Yes, No), the zone of the dose administration (I, II, III, IV, V, VI) and "Was the total volume of dose administered per protocol?" (Yes, No). In addition, the volume of study drug administered (continuous variable) will be summarized in minutes using summary statistics.

## 10.2 Adverse Events

All adverse event summaries will be restricted to Treatment Emergent Adverse Events (TEAE), which are defined as those AEs that occurred after dosing and those existing AEs that worsened during the study. Verbatim terms on case report forms will be mapped to preferred terms and system organ classes using the MedDRA dictionary (version 9.1).

Each adverse event summary will be displayed by dose cohort. Summaries that are displayed by system organ class and preferred terms will be ordered by descending order of incidence of system organ class and preferred term within each system organ class. Summaries of the following types will be presented:

- Subject incidence of TEAEs and total number of unique TEAEs by MedDRA system organ class and preferred term;
- Subject incidence of TEAEs by MedDRA system organ class, preferred term, and highest severity. At each level of subject summarization a subject is classified according to the highest severity if the subject reported one or more events. AEs with missing severity will be considered severe for this summary;

- Subject incidence of TEAEs by MedDRA system organ class, preferred term, and closest relationship to study drug (Related/Not Related). At each level of subject summarization a subject is classified according to the closest relationship if the subject reported one or more events. AEs with a missing relationship will be considered related for this summary;
- Subject incidence of serious TEAEs and total number of unique serious TEAEs by MedDRA system organ class and preferred term.

## 10.3 Clinical Laboratory Evaluation

Before the first dose of medication and at Day 15 (Pre-Dose), Day 16, Day 28, Day 59, Day 91, Day 180 and Day 365 of the study, clinical laboratory evaluations (Hematology, Chemistry, Urinalysis) will be taken. Laboratory parameters will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized. Baseline is defined as the last non-missing value prior to first dose of study drug.

In addition, shift tables (i.e., low-normal-high at baseline versus low-normal-high at follow-up in a 3-by-3 contingency table) will be provided to assess changes in laboratory values from baseline to most abnormal follow-up result.

## 10.4 Physical Examinations

At Screening, a physical examination will be carried out on the following body systems: HEENT, Skin/Dermatologic, Lymph Nodes, Chest/Lungs, Heart/Cardiovascular, Abdomen, Extremities, Neurologic, Stool for Occult Blood, Other. Assessments for each of the body systems will be one of the following: Normal, Abnormal-Not Clinically Significant, Abnormal-Clinically Significant, Not Done. At Day 15 (Pre-Dose), Day 28, Day 59, Day 91, Day 180 and Day 365, changes in any of the body systems will be recorded.

Shift tables will be provided to assess changes in body systems from baseline to each follow up visit.

## 10.5 Vital Signs

At each visit, vital signs will be collected. Additional vital signs will be collected on the days of dosing (Day 1 and Day 15) at 15, 30 and 60 minutes post dose. Vital signs will be summarized using descriptive statistics at baseline and at each post baseline time point.

Changes from baseline will also be summarized. Baseline is defined as the last non-missing value prior to first dose of study drug.

## 10.6 Retinal Fundoscopy

A retinal fundoscopy of each eye will be performed at Screening and at Day 365. Each eye will be given one of the following assignments: Normal, Abnormal-Not Clinically Significant, Abnormal-Clinically Significant. Shift tables will be provided to assess changes in retinal fundoscopy.

## 10.7 Infection Tests

Tests will be carried out to determine the presence of selected infections at Screening and on Day 59, Day 180 and Day 365. Infections to be tested will include Hepatitis BSAg, HCV, HTLV, CMV and VDRL. The counts and percentages of number of subjects reporting a positive infection test will be presented by visit and infection type.

## 10.8 Tumor Marker

Measurements of selected tumor markers will be made at Screening, Day 59, Day 180 and Day 365. Tumor markers to be considered are the following: Alpha Fetoprotein (AFP), Carcino Embryonic Antigen (CEA), Prostate Specific Antigen (PSA), Cancer Antigen 19-9 (CA19-9), CA 125. Tumor marker results will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized.

## 10.9 Injection Site Reaction

Assessments of the existence of an injection site reaction are planned for Day 1 (Post-Dose), Day 8, Day 15 (Post-Dose), Day 16, Day 21, Day 28 and Day 59. The number and percentage of subjects with an injection site reaction will be summarized.

## 10.10 Prior and Concomitant Medications

Verbatim terms on case report forms will be mapped to Anatomical/Therapeutic/Chemical (ATC) Level 4 categories and Drug Reference Names using the World Heath Organization (WHO) dictionary (version 5.3).

Prior medications are those medications taken within 30 days prior to the initial dose of study drug. Concomitant medications are those medications taken after the initial dose of study drug. Prior and concomitant medications will be summarized for each treatment by

WHO ATC class and medication name. These summaries will present the number and percentage of subjects using each medication. Subjects may have more than one medication per ATC category and medication. At each level of subject summarization, a subject is counted once if he/she reported one or more medications at that level. Each summary will be ordered by descending order of incidence of ATC class and medication within each ATC class.

## 11. PHARMACOKINETICS

VM202 DNA levels will be determined before dose on Day 1. In addition, VM202 DNA levels will be collected on Day 21 and Day 59 (if DNA is detected on Day 21). VM202 DNA level results will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized.

## 12. PHARMACODYNAMICS

An endothelial progenitor cell assay test will be performed at Screening, Day 1 (Post Dose), Day 15 (Post Dose), Day 28, Day 59, Day 180 and Day 365. Endothelial progenitor cell assay test results will be summarized using descriptive statistics at baseline and at each post baseline time point. Changes from baseline will also be summarized.

Serum HGF levels will be collected at Day 1 (Pre-Dose), Day 8, Day 15 (Pre-Dose), Day 21 and Day 59. Results and changes from baseline will be presented by time point.

Anti-HGF antibodies data will be collected on Day 1 (Pre-Dose), Day 15 (Pre-Dose), Day 59 and possibly Day 180. Results will be presented in listings.

# APPENDIX A: LIST OF TABLES AND LISTINGS

## List of Tables

| Table | |
|---|---|
| Number | Table Description |
| 1 | Subject Disposition |
| 2 | Demographic Characteristics (ITT/Safety Population) |
| 3 | Abnormal Medical History at Baseline (Safety Population) |
| 4 | Peripheral Vascular Disease Intervention History (Safety Population) |
| 5 | Ulcer Measurement (ITT Population) |
| 6 | Ankle Brachial-Index (ITT Population) |
| 7 | Toe Brachial-Index (ITT Population) |
| 8 | Visual Analogue Scale for Pain (ITT Population) |
| 9 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> (ITT Population) |
| 10 | Subject Analgesic Use (ITT Population) |
| 11 | Study Drug Exposure(Safety Population) |
| 12 | Treatment Emergent Adverse Events by Cohort (Safety Population) |
| 13 | Treatment Emergent Adverse Events by System Organ Class and Severity |
| | (Safety Population) |
| 14 | Treatment Emergent Adverse Events by System Organ Class and |
| | Relationship to Study (Safety Population) |
| 15 | Treatment Emergent Serious Adverse Events by Cohort (Safety |
| | Population) |
| 16.1 | Hematology (Safety Population) |
| 16.2 | Chemistry (Safety Population) |
| 16.3 | Urinalysis (Safety Population) |
| 17.1 | Hematology – Shift from Baseline (Safety Population) |
| 17.2 | Chemistry – Shift from Baseline (Safety Population) |
| 17.3 | Urinalysis – Shift from Baseline (Safety Population) |
| 18 | Physical Examinations- Shift from Baseline (Safety Population) |
| 19 | Vital Signs (Safety Population) |
| 20 | Retinal Fundoscopy- Shift from Baseline (Safety Population) |
| 21 22 | Infection Tests (Safety Population) |
| | Tumor Markers (Safety Population) |
| 23 | Injection Site Reaction (Safety Population) |
| 24 | Concomitant Medications (Safety Population) |

# List of Tables (cont)

| Table | |
|--------|----------------------------------------------------|
| Number | Table Description |
| 25 | VM202 DNA Levels (ITT Population) |
| 26 | Endothelial Progenitor Cell Assay (ITT Population) |
| 27 | Serum HGF Levels (ITT Population) |

# List of Data Listings

| Listing | | CRF |
|---|---|---|
| Number | Listing Description | Plate(s) |
| 1 | Subject Disposition (including Informed Consent | Derived,1, |
| | Date/Investigator Signature) | 100 |
| 2 | Inclusion/ Exclusion Criteria | 1-3 |
| 3 | Demographics/ 12-Lead ECG Results | 4,9 |
| 4 | Medical History | 5 |
| 5 | Peripheral Vascular Disease Intervention History | 6 |
| 6 | Serum/Urine Pregnancy Test/ Mammogram/ Pap Smear | 4,15,19,24 |
| | Results/ Pregnancy Outcome | |
| 7 | Ulcer Measurements | 16 |
| 8 | High Resolution MRA/ Injection Site Reaction | 16 |
| 9 | Assessment of CLI | 17 |
| 10 | Hemodynamic Assessments | 18 |
| 11 | Visual Analogue Scale for Pain | 19 |
| 12 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> | 19 |
| 13 | Concomitant Medications Identified as being Analgesic in | 98 |
| | Nature | |
| 14 | Study Drug Administration | 20 |
| 15 | Adverse Events | 97 |
| 16 | Serious Adverse Events | 97 |
| 17 | Hematology | 11 |
| 18 | Chemistry | 12 |
| 19 | Urinalysis | 13 |
| 20 | Physical Examinations | 7,8 |
| 21 | Vital Signs | 9 |
| 22 | Retinal Fundoscopy/ Chest X-Ray/ CT Scan | 10 |
| 23 | Infection Tests | 14 |
| 24 | Tumor Markers | 15 |
| 25 | Concomitant Medications | 98 |
| 26 | VM202 DNA Levels (include Collection Date/Time from CRF) | 16, Lab |
| 27 | Endothelial Progenitor Cell Assay | 14 |
| 28 | Serum HGF/ Anti HGF Antibodies (include Collection | 14, Lab |
| | Date/Time from CRF) | |
| 29 | Telephone Follow-Up Contact | 22 |
| 30 | Waiver | 23 |

# List of Data Listings (cont)

| Listing | | CRF |
|---------|---------------------|----------|
| Number | Listing Description | Plate(s) |
| 31 | Death | 101 |

# APPENDIX B: TABLE LAYOUTS

Viromed Co., Ltd. Page 1 of x Protocol Number: US-06-1-001

Table 1 **Subject Disposition** All Subjects

| | VM202- 2 mg | VM202- 4 mg | VM202-8 mg | VM202- 16 mg |
|---|---|---|---|---|
| Subjects Enrolled | n | n | n | n |
| Safety Population [1] | n | n | n | n |
| ITT Population [2] | n | n | n | n |
| Received 2 Doses of VM202? | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) |
| Last Visit Completed | | | | |
| Any Visit Prior to Visit- Day 21 | n (%) | n (%) | n (%) | n (%) |
| Visit- Day 21 | n (%) | n (%) | n (%) | n (%) |
| Visit- Day 28 | n (%) | n (%) | n (%) | n (%) |
| Visit- Day 59 | n (%) | n (%) | n (%) | n (%) |
| Visit- Day 91 | n (%) | n (%) | n (%) | n (%) |
| Visit- Day 180 | n (%) | n (%) | n (%) | n (%) |
| Visit- Day 365 | n (%) | n (%) | n (%) | n (%) |
| Completed Study? | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) |
| Primary Reason for Discontinuation | | | | |
| Screen failure | n (%) | n (%) | n (%) | n (%) |
| Lost to Follow-up | n (%) | n (%) | n (%) | n (%) |
| Adverse Event | n (%) | n (%) | n (%) | n (%) |
| Non-compliance | n (%) | n (%) | n (%) | n (%) |
| Subject withdrew consent | n (%) | n (%) | n (%) | n (%) |
| Principal Investigator decision | n (%) | n (%) | n (%) | n (%) |
| Subject requires intervention for treatment of acute limb ischemia | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) |

<sup>\*</sup> Percentages based on number of subjects Enrolled.
[1] All subjects who received at least one dose of study drug.

<sup>[2]</sup> All subjects who received at least one dose of study drug and had at least one post dose assessment.

Table 2
Demographic Characteristics
ITT Population

| | VM202- 2 mg<br>(N= ) | VM202- 4 mg<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|---|
| Age (years) [1] | | | | |
| N | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Sex | | | | |
| Male | n (%) | n (%) | n (%) | n (%) |
| Female | n (%) | n (%) | n (%) | n (%) |
| Ethnicity | | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) | n (%) |
| Race | | | | |
| American Indian or Alaska Native | n (%) | n (%) | n (%) | n (%) |
| Asian | n (%) | n (%) | n (%) | n (%) |
| Black or African American | n (%) | n (%) | n (%) | n (%) |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) | n (%) |
| White | n (%) | n (%) | n (%) | n (%) |
| Multiple Races Checked | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Age calculated by determining the number of years between the date of informed consent and the date of birth. path\t program.sas date time

Programmer note Table 2.2 will be identical to Table 2.1 for the Safety Population.

Table 3 Abnormal Medical History at Baseline Safety Population

| De de Contant | VM202- 2 mg | VM202- 4 mg | VM202- 8 mg | VM202- 16 mg |
|---|---|---|---|---|
| Body System | (N= ) | (N= ) | (N= ) | (N= ) |
| Respiratory | n (%) | n (%) | n (%) | n (%) |
| Cardiovascular | n (%) | n (%) | n (%) | n (%) |
| Gastrointestinal | n (%) | n (%) | n (%) | n (%) |
| Hepatic | n (%) | n (%) | n (%) | n (%) |
| Endocrine/Metabolic | n (%) | n (%) | n (%) | n (%) |
| Central Nervous System | n (%) | n (%) | n (%) | n (%) |
| Hematopoietic/Lymphatic | n (%) | n (%) | n (%) | n (%) |
| Dermatological | n (%) | n (%) | n (%) | n (%) |
| Musculoskeletal | n (%) | n (%) | n (%) | n (%) |
| Genitourinary/Reproductive | n (%) | n (%) | n (%) | n (%) |
| Psychiatric | n (%) | n (%) | n (%) | n (%) |
| Alcohol/Drug Abuse | n (%) | n (%) | n (%) | n (%) |
| Drug Allergy | n (%) | n (%) | n (%) | n (%) |
| Non-Drug Allergy | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) |

Table 4
Peripheral Vascular Disease Intervention
Safety Population

| Intervention | VM202- 2 mg<br>(N= ) | VM202- 4 mg<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|---|
| merventon | (11- ) | (11- ) | (11- ) | (11- ) |
| PTA | n (%) | n (%) | n (%) | n (%) |
| Peripheral bypass | n (%) | n (%) | n (%) | n (%) |
| Amputation above the knee | n (%) | n (%) | n (%) | n (%) |
| Amputation below the knee | n (%) | n (%) | n (%) | n (%) |
| Atherectomy | n (%) | n (%) | n (%) | n (%) |
| Surgical bypass | n (%) | n (%) | n (%) | n (%) |
| Endarterectomy | n (%) | n (%) | n (%) | n (%) |
| Thrombectomy | n (%) | n (%) | n (%) | n (%) |
| Stent placement | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) |

Page 1 of x

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 5 Ulcer Measurement (cm<sup>2</sup>) [1] ITT Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 | mg (N= ) | VM202-10 | 5 mg (N= ) |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [3] | Result | Change [3] | Result | Change [3] | Result | Change [3] |
| Baseline [2] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | XX, XX | | xx, xx | |
| Day 15 (Pre-Dose) | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX |
| Day 28 | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX |
| Day 59 | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |

path\t\_program.sas date time

Programmer Note Repeat for all available time points.

<sup>[1]</sup> Measurement taken was the largest contiguous area of ulceration.[2] Baseline defined as measurement taken most closely prior to first study drug administration.

<sup>[3]</sup> Change= Change from Baseline

Viromed Co., Ltd. Page 1 of x Protocol Number: US-06-1-001

> Table 6 Ankle Brachial-Index (mmHg) ITT Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 | mg (N= ) | VM202-10 | 6 mg (N= ) |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Index Limb | | | | | | | | |
| Right | n (%) | | n (%) | | n (%) | | n (%) | |
| Left | n (%) | | n (%) | | n (%) | | n (%) | |
| Delt | П (70) | | 11 (70) | | 11 (70) | | 11 (70) | |
| ABI Index Leg | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| , | , | | , | | , | | , | |
| Day 15 (Pre-Dose) | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x | XX.X | xx.x | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| ABI Non-Index Leg | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| , | , | | , | | , | | , | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.
[2] Change= Change from Baseline

Viromed Co., Ltd. Page 1 of x

Protocol Number: US-06-1-001

Table 7 Toe Brachial-Index (mmHg) ITT Population

| | VM202-2 | mg (N= ) | VM202- 4 mg (N= ) | | VM202-8 | mg (N= ) | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| TBI Index Toe | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | | XX, XX | |
| Day 15 (Pre-Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |
| TBI Non-Index Toe | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | | xx, xx | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note For each measurement, repeat for all available time points.

<sup>[2]</sup> Change= Change from Baseline

Table 8 Visual Analogue Scale for Pain (mm) ITT Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 | mg (N= ) | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | | xx, xx | |
| Day 15 (Pre-Dose) | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX |
| Day 28 | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Day 59 | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note Repeat for all available time points.

<sup>[2]</sup> Change= Change from Baseline

Table 9
Transcutaneous Oxygen Pressure Assessment- TcPO<sub>2</sub> (mmHg)
ITT Population

| | VM202-2 | VM202- 2 mg (N= ) | | mg (N= ) | VM202-8 | mg (N= ) | VM202-16 mg (N= | |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Anterior Calf | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | XX, XX | | XX, XX | |
| Day 15 (Pre-Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |
| Posterior Calf | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | | xx, xx | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note For each measurement, repeat for all available time points. Results for other measurements to be shown include Dosrum Foot and Chest..

<sup>[2]</sup> Change= Change from Baseline

Protocol Number: US-06-1-001

Table 10 Subject Analgesic Use [1] ITT Population

| | VM202- 2 mg<br>(N= ) | VM202- 4 mg<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|---|
| Subject reported using analgesic d | uring study? | | | |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) |

[1] Subject identified as having used analgesic based on whether subject reported using any concomitant medications considered to be an analgesic.

path\t\_program.sas date time

Programmer Note:

Table 11 Study Drug Exposure Safety Population

| | VM202- 2 mg | VM202- 4 mg | VM202-8 mg | VM202- 16 mg |
|---|---|---|---|---|
| | (N= ) | (N= ) | (N= ) | (N= ) |
| Day 1 Dose Administered? | | | | |
| | - (0/) | - (0/) | - (0/) | - (0/) |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No, DLT from previous injection | n (%) | n (%) | n (%) | n (%) |
| No, Other | n (%) | n (%) | n (%) | n (%) |
| Zone of Injections | | | | |
| I | n (%) | n (%) | n (%) | n (%) |
| П | n (%) | n (%) | n (%) | n (%) |
| Ш | n (%) | n (%) | n (%) | n (%) |
| IV | n (%) | n (%) | n (%) | n (%) |
| V | n (%) | n (%) | n (%) | n (%) |
| VI | n (%) | n (%) | n (%) | n (%) |
| Total Volume Administered per Protocol? | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) |
| Time Dose Administration (mg) | | | | |
| N | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 15 | | | | |
| Dose Administered? | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) |
| 110 | 11 (70) | 11 (70) | 11 (70) | 11 (70) |

Page 1 of x

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 12 Treatment Emergent Adverse Events by Cohort [1] Safety Population

| | VM202- 2 mg (N= ) | | VM202- 4 mg (N= ) | | VM202-8 mg (N= ) | | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| | Number of | Number of | Number of | Number of | Number of | Number of | Number of | Number of |
| System Organ Class / Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Adverse Event | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| • | | | | | | | | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |

[1] At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.

Protocol Number: US-06-1-001

Table 13
Treatment Emergent Adverse Events by System Organ Class and Severity [1]
Safety Population
Part 1 of 2

| | VM202- 2 mg (N= ) | | | | | VM202-4 mg (N= ) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Mild | Moderate | Severe | Life Threat. | Death | Mild | Moderate | Severe | Life Threat. | Death |
| Subjects Reporting at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| - | | | | | | | | | | |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the highest severity.

Protocol Number: US-06-1-001

Table 13
Treatment Emergent Adverse Events by System Organ Class and Severity [1]
Safety Population
Part 2 of 2

| | VM202-8 mg (N= ) | | | | | VM202- 16 mg (N= ) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Mild | Moderate | Severe | Life Threat. | Death | Mild | Moderate | Severe | Life Threat. | Death |
| Subjects Reporting at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| • | | | | | | | | | | |
| • | | | | | | | | | | |
| System Organ Class 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the highest severity.

Protocol Number: US-06-1-001

Table 14
Treatment Emergent Adverse Events by System Organ Class and Relationship to Study Drug [1]
Safety Population

| | VM202- 2 mg (N= ) | | VM202- 4 mg (N= ) | | VM202-8 mg (N= ) | | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Related [2] | Not Related [3] | Related [2] | Not Related [3] | Related [2] | Not Related [3] | Related [2] | Not Related [3] |
| Subjects Reporting at Least One Adverse Event | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| - | | | | | | | | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the closest relationship to study drug.

<sup>[2]</sup> Includes all events reported as "Possibly," "Probably," or of "Definitely" relationship to study drug.

<sup>[3]</sup> Includes all events reported as "Unlikely" or "Unrelated" relationship to study drug.

Protocol Number: US-06-1-001

Table 15 Treatment Emergent Serious Adverse Events by Cohort [1] Safety Population

| | VM202- 2 mg (N= ) | | VM202- 4 mg (N= ) | | VM202-8 mg (N= ) | | VM202- 16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| | Number of | Number of | Number of | Number of | Number of | Number of | Number of | Number of |
| System Organ Class / Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Serious Adverse Event | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| - | | | | | | | | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.
Protocol Number: US-06-1-001

Table 16.1 Hematology Safety Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 | mg (N= ) | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| Analyte | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Analyte #1 (unit) | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | XX.X | | xx.x | | xx.x | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | | xx, xx | |
| Day 15 (Pre-Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 16 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX |
| Day 28 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note Repeat for all available time points and analytes. Analytes to be shown include Hematocrit, Hemoglobin, RBC, WBC, Platelets, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, MCV, MCHC, MCH.

<sup>[2]</sup> Change= Change from Baseline

Table 16.2 Chemistry Safety Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 | mg (N= ) | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| Analyte | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Analyte #1 (unit) | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| Day 15 (Pre-Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Day 16 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Day 28 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

Protocol Number: US-06-1-001

path\t\_program.sas date time

Programmer Note Repeat for all available time points and analytes. Analytes to be shown include Albumin, Alkaline Phosphate, ALT, AST, Bicarbonate, BUN, Calcium, Chloride, Creatinine, GGT Glucose, LDH, Phosphorus, Sodium, Total Bilirubin, Total Protein, Uric Acid.

<sup>[2]</sup> Change= Change from Baseline

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 16.3 Urinalysis Safety Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 | mg (N= ) | VM202- 16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| Analyte | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Analyte #1 (unit) | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | | xx, xx | |
| Day 15 (Pre-Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Day 16 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Day 28 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note Repeat for all available time points and analytes. Analytes to be shown include Specific Gravity, pH.

<sup>[2]</sup> Change= Change from Baseline

Viromed Co., Ltd. Page 1 of x Protocol Number: US-06-1-001

Table 17 1

| Table 17.1 |
|---------------------------------|
| Hematology- Shift from Baseline |
| Safety Population |

| VM202- 16 mg (N= ) |
|--------------------|
| High Normal Low |
| n (%) n (%) n (%) |
| n (%) n (%) n (%) |
| n (%) n (%) n (%) |
| n (%) n (%) n (%) |
| n (%) n (%) n (%) |
| n (%) n (%) n (%) |
| n (%) n (%) |

path\t\_program.sas date time

Programmer Note If a subject has both a High and Low post dose result, the subject will be assigned a High result for the Most Abnormal Post Dose Result,. Analytes to be shown include Hematocrit, Hemoglobin, RBC, WBC, Platelets, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, MCV, MCHC, MCH.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

<sup>[2]</sup> Follow Up defined as most abnormal post dose result.

Viromed Co., Ltd. Page 1 of x Protocol Number: US-06-1-001

T-11- 47 0

| Table 17.2 |
|--------------------------------|
| Chemistry- Shift from Baseline |
| Safety Population |

| Baseline [1] | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| VM202- 2 mg (N= ) | | | VM | VM202-4 mg (N=) | | | VM202-8 mg (N=) | | | VM202-16 mg (N=) | |
| High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low |
| n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | | n (%) | n (%) | | n (%) | n (%) | | n (%) | n (%) | n (%) |
| n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | | n (%) | n (%) | | n (%) | n (%) | | n (%) | n (%) | n (%) |
| n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) n (%) n (%) n (%) n (%) | High Normal n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) | High Normal Low | High Normal Low High | High Normal Low High Normal | VM202- 2 mg (N= ) VM202- 4 mg (N= ) High Normal Low High Normal Low n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) | VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM High Normal Low High Normal Low High n (%) n (%) n (%) n (%) n ( | VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) High Normal Low High Normal Low High Normal n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) <t< td=""><td>VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) High Normal Low High Normal Low High Normal Low n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) <td< td=""><td>VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) VM2 High Normal Low High Normal Low High n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n</td><td>VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) VM202- 16 mg (1 High Normal Low High Normal Low High Normal Low High Normal n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%)</td></td<></td></t<> | VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) High Normal Low High Normal Low High Normal Low n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) <td< td=""><td>VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) VM2 High Normal Low High Normal Low High n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n</td><td>VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) VM202- 16 mg (1 High Normal Low High Normal Low High Normal Low High Normal n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%)</td></td<> | VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) VM2 High Normal Low High Normal Low High n (%) n | VM202- 2 mg (N= ) VM202- 4 mg (N= ) VM202- 8 mg (N= ) VM202- 16 mg (1 High Normal Low High Normal Low High Normal Low High Normal n (%) n (%) |

path\t\_program.sas date time

Programmer Note If a subject has both a High and Low post dose result, the subject will be assigned a High result for the Most Abnormal Post Dose Result. Analytes to be shown include Albumin, Alkaline Phosphate, ALT, AST, Bicarbonate, BUN, Calcium, Chloride, Creatinine, GGT Glucose, LDH, Phosphorus, Sodium, Total Bilirubin, Total Protein, Uric Acid.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

<sup>[2]</sup> Follow Up defined as most abnormal post dose result.

Protocol Number: US-06-1-001

## Table 17.3 Urinalysis- Shift from Baseline Safety Population

| | | | | | | Basel | ine [1] | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | VM | VM202- 2 mg (N= ) | | VM | VM202-4 mg (N=) | | | VM202-8 mg (N= ) | | | VM202- 16 mg (N= ) | |
| Follow Up [2] | High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low |
| Analyte #1 (unit) | | | | | | | | | | | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Analyte #2 (unit) | | | | | | | | | | | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note If a subject has both a High and Low post dose result, the subject will be assigned a High result for the Most Abnormal Post Dose Result. Analytes to be shown include Specific Gravity, pH.

<sup>[2]</sup> Follow Up defined as most abnormal post dose result.

Protocol Number: US-06-1-001

## Table 18 Physical Examinations- Shift from Baseline Safety Population

Screening Visit

| | Set Colling Visit | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | VM | 202- 2 mg (N | = ) | VM | 202- 4 mg (N | = ) | VM | 202-8 mg (N | <b>=</b> ) | VM: | 1= ) | |
| | | Abn, Not | Abn, | | Abn, Not | Abn, | | Abn, Not | Abn, | | Abn, Not | Abn, |
| Body System | Normal | CS[1] | CS [2] | Normal | CS[1] | CS [2] | Normal | CS[1] | CS [2] | Normal | CS[1] | CS [2] |
| Body System #1 | | | | | | | | | | | | |
| Day 15 | n | | | n | | | n | | | n | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 28 | n | | | n | | | n | | | n | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 59 | n | | | n | | | n | | | n | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Programmer Note Repeat for all available time points and body systems. Body Systems to be shown include HEENT, Skin/Dermatologic, Lymph Nodes, Chest/Lungs, Heart/Cardiovascular, Abdomen, Extremities, Neurologic, Stool for Occult Blood, Other.

<sup>[1]</sup> Abn, Not CS= Abnormal, Not Clinically Significant

<sup>[2]</sup> Abn, CS= Abnormal, Clinically Significant

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 19 Vital Signs Safety Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 | mg (N= ) | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| Vital Sign | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| T (D ( 4 ) | | | | | | | | |
| Heart Rate (bpm) | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N<br>(GD) | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| Day 1 (15 Minutes Post Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Day 1 (30 Minutes Post Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX |
| Day 1 (60 Minutes Post Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| , | , | , | , | , | , | , | , | , |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.
[2] Change= Change from Baseline

path\t\_program.sas date time

Programmer Note Repeat for all available time points and vital signs.

Protocol Number: US-06-1-001

Table 20 Retinal Fundoscopy- Shift from Baseline Safety Population

| | | Screening/Baseline | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | VM | 202-2 mg (N | = ) | VM | 202- 4 mg (N | = ) | VM202- 8 mg (N= ) | | | VM202- 16 mg (N= ) | | |
| | | Abn, Not | Abn, | | Abn, Not Abn, | | | Abn, Not Abn, | | | Abn, Not | Abn, |
| | Normal | CS[1] | CS [2] | Normal | CS[1] | CS [2] | Normal | CS[1] | CS [2] | Normal | CS[1] | CS [2] |
| Day 365/ Early Termination | | | | | | | | | | | | |
| Right | | | | | | | | | | | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Left | | | | | | | | | | | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Abn, Not CS= Abnormal, Not Clinically Significant [2] Abn, CS= Abnormal, Clinically Significant

path\t\_program.sas date time

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 21 Infection Tests Safety Population

| | VM | 202- 2 mg ( | (N= ) | VM | 202- 4 mg ( | N= ) | VM | 202- 8 mg ( | N= ) | VM202- 16 mg (N= ) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pos | Neg | Not Done | Pos | Neg | Not Done | Pos | Neg | Not Done | Pos | Neg | Not Done |
| Screening | n | | | n | | | n | | | n | | |
| Hepatitis BSAg | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HCV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HTLV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| CMV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| VDRL | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 59 | n | | | n | | | n | | | n | | |
| Hepatitis BSAg | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HCV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HTLV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| CMV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| VDRL | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 180 | n | | | n | | | n | | | n | | |
| Hepatitis BSAg | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HCV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HTLV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| CMV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| VDRL | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 365 | n | | | n | | | n | | | n | | |
| Hepatitis BSAg | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HCV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HTLV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| CMV | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| VDRL | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| ·DILL | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) |

path\t\_program.sas date time

Table 22 Tumor Markers Safety Population

| | VM202- 2 | mg (N= ) | VM202-4 | mg (N= ) | VM202-8 mg (N= ) | | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| Tumor Marker | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| AFP (Alpha Fetoprotein) (ng/mL)<br>Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | XX, XX | | XX, XX | |
| Day 15 (Pre-Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 59 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX |
| Day 180 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x | xx.x | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

Protocol Number: US-06-1-001

path\t\_program.sas date time

Programmer Note Repeat for all available time points and tumor markers. Tumor Markers to be shown include CEA (Carcino Embryonic Antigen), PSA (Prostate Specific Antigen), CA 19-9 (Cancer Antigen 19-9), CA 125..

<sup>[2]</sup> Change= Change from Baseline

Viromed Co., Ltd. Page 1 of x

Viromed Co., Ltd. Protocol Number: US-06-1-001

## Table 23 Injection Site Reaction Safety Population

| | VM202- 2 mg<br>(N= ) | VM202- 4 mg<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|---|
| Subject reported an Injection Site | Reaction? | | | |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Programmer Note:

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 24 Concomitant Medications [1] Safety Population

| ATC Drug Class / Medication Term | VM202- 2 mg | VM202- 4 mg | VM202- 8 mg | VM202- 16 mg |
|---|---|---|---|---|
| | (N= ) | (N= ) | (N= ) | (N= ) |
| Subjects Receiving any Concomitant Medications | n (%) | n (%) | n (%) | n (%) |
| Drug Class 1 Medication Term 1 Medication Term 2 . | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) |
| Drug Class 2 Medication Term 1 Medication Term 2 | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) |

[1] At each level of summation (overall, ATC drug class, medication term), subjects reporting more than medication are counted only once.

path\t\_program.sas date time

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 25 VM202 DNA Levels (unit) ITT Population

| | VM202- 2 mg (N= ) | | VM202- 4 mg (N= ) | | VM202-8 mg (N= ) | | VM202-16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| Day 21 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 59 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note Repeat for all available time points.

<sup>[2]</sup> Change= Change from Baseline

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 26 Endothelial Progenitor Cell Assay (%) ITT Population

| | VM202- 2 | VM202- 2 mg (N= ) | | VM202- 4 mg (N= ) | | VM202-8 mg (N= ) | | VM202-16 mg (N= ) |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | | xx, xx | |
| Day 1 (Post Dose) | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Day 15 (Post Dose) | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Day 28 | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note Repeat for all available time points.

<sup>[2]</sup> Change= Change from Baseline

Viromed Co., Ltd. Protocol Number: US-06-1-001

Table 27 Serum HGF Levels (unit) ITT Population

| | VM202-2 mg (N=) | | VM202- 4 mg (N= ) | | VM202-8 mg (N= ) | | VM202- 16 mg (N= ) | |
|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| - E 50 | | | | | | | | |
| Baseline [1] | | | | | | | | |
| N | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| Day 8 | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 15 (Pre-Dose) | | | | | | | | |
| Ň | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 21 | | | | | | | | |
| N | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | | | | | | | |
| IVIIII, IVIAA | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note Repeat for all available time points.

<sup>[2]</sup> Change= Change from Baseline